CLINICAL TRIAL: NCT06277336
Title: Effects of Intravenous [Pyr1]Apelin-13 on Healthy Volunteers With Artificially Induced SIAD- the ESCAPE Study
Brief Title: Effects of Intravenous [Pyr1]Apelin-13 on Healthy Volunteers With Artificially Induced SIAD
Acronym: ESCAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-01716; kt23ChristCrain3
Record Dates: First submitted 2024-01-30; First posted 2024-02-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: SIAD - Syndrome of Inappropriate Antidiuresis; Hyponatremia
Keywords: Apelin
MeSH Terms: conditions — Inappropriate ADH Syndrome; Hyponatremia | interventions — Apelin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Healthy Volunteers Intervention Order: Placebo, Apelin Low Dose, Apelin High Dose (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Healthy Volunteers Healthy Patients Intervention Order: Apelin Low Dose, Apelin High Dose, Placebo (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Healthy Volunteers Intervention Order: Apelin High Dose, Placebo, Apelin Low Dose (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Healthy Volunteers Intervention Order: Placebo, Apelin High Dose, Apelin Low Dose (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Healthy Volunteers Intervention Order: Apelin Low Dose, Placebo, Apelin High Dose (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Healthy Volunteers Intervention Order: Apelin High Dose, Apelin Low Dose, Placebo (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Artificial SIAD induction (water loading and desmopressin administration) is performed.
  Interventions: Drug: Placebo; Drug: Apelin Low Dose; Drug: Apelin High Dose
- Chronic SIAD Patients Intervention Order: Placebo, Selected Apelin Dose (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Interventions: Drug: Placebo; Drug: Selected Apelin Dose
- Chronic SIAD Patients Intervention Order: Selected Apelin Dose, Placebo (Experimental): The intervention sequence is assigned in random order. Each intervention corresponds to a visit of 11h. A wash-out period of 2 to 8 weeks is planned between interventions.
  Interventions: Drug: Placebo; Drug: Selected Apelin Dose

INTERVENTIONS:
Drug: Placebo — Artificial SIAD induction:
  * Oral water intake of 30ml/kg body weight in one hour (timepoint -2 to timepoint -1)
  * Intravenous bolus of desmopressin 4 μg i.v. (Minirin®, Ferring AG) (timepoint -1)
  * 300ml NaCl 0.45% (B. Braun Medical AG) over 1 hour (timepoint -1 to 0)
  Study infusion (timepoint 0 to timepoint +3):
  * 180-ml NaCl 0.45% infusion (placebo) over 3 hours (60ml per h)
Drug: Apelin Low Dose — Artificial SIAD induction:
  * Oral water intake of 30ml/kg body weight in one hour (timepoint -2 to timepoint -1)
  * Intravenous bolus of desmopressin 4 μg i.v. (Minirin®, Ferring AG) (timepoint -1)
  * 300ml NaCl 0.45% (B. Braun Medical AG) over 1 hour (timepoint -1 to 0)
  Study infusion (timepoint 0 to timepoint +3):
  * 180-ml infusion of [Pyr1]apelin-13 in NaCl 0.45% over 3 hours at an infusion rate of 1 nmol/min (60ml per h)
  Arms: Healthy Volunteers Healthy Patients Intervention Order: Apelin Low Dose, Apelin High Dose, Placebo; Healthy Volunteers Intervention Order: Apelin High Dose, Apelin Low Dose, Placebo; Healthy Volunteers Intervention Order: Apelin High Dose, Placebo, Apelin Low Dose; Healthy Volunteers Intervention Order: Apelin Low Dose, Placebo, Apelin High Dose; Healthy Volunteers Intervention Order: Placebo, Apelin High Dose, Apelin Low Dose; Healthy Volunteers Intervention Order: Placebo, Apelin Low Dose, Apelin High Dose
Drug: Apelin High Dose — Artificial SIAD induction:
  * Oral water intake of 30ml/kg body weight in one hour (timepoint -2 to timepoint -1)
  * Intravenous bolus of desmopressin 4 μg i.v. (Minirin®, Ferring AG) (timepoint -1)
  * 300ml NaCl 0.45% (B. Braun Medical AG) over 1 hour (timepoint -1 to 0)
  Study infusion (timepoint 0 to timepoint +3):
  * 180-ml infusion of [Pyr1]apelin-13 in NaCl 0.45% over 3 hours at an infusion rate of 10 nmol/min (60ml per h)
  Arms: Healthy Volunteers Healthy Patients Intervention Order: Apelin Low Dose, Apelin High Dose, Placebo; Healthy Volunteers Intervention Order: Apelin High Dose, Apelin Low Dose, Placebo; Healthy Volunteers Intervention Order: Apelin High Dose, Placebo, Apelin Low Dose; Healthy Volunteers Intervention Order: Apelin Low Dose, Placebo, Apelin High Dose; Healthy Volunteers Intervention Order: Placebo, Apelin High Dose, Apelin Low Dose; Healthy Volunteers Intervention Order: Placebo, Apelin Low Dose, Apelin High Dose
Drug: Selected Apelin Dose — Study infusions (timepoint 0 to timepoint +3):
  * 180-ml NaCl 0.45% infusion (placebo) over 3 hours (60ml per h)
  * 180-ml infusion of [Pyr1]apelin-13 in NaCl 0.45% over 3 hours based on the best performing apelin dose (from Low Dose or High Dose) in healthy volunteers corresponding to one of the following options:
    1. at an infusion rate of 1 nmol/min (60ml per h) OR
    2. at an infusion rate of 10 nmol/min (60ml per h)
  In case both apelin dosis performed equally well in the healthy volunteers population the lower dose will be selected.
  Arms: Chronic SIAD Patients Intervention Order: Placebo, Selected Apelin Dose; Chronic SIAD Patients Intervention Order: Selected Apelin Dose, Placebo

SUMMARY:
Hyponatremia is a common electrolyte imbalance which often results from hormonal disregulation. The study aims to investigate whether the apelin hormone, which plays a role in regulating salt and water balance in the body, can be used to treat hyponatremia.

The study will involve healthy volunteers who will be given a medication that causes their bodies to retain water, thus inducing a temporary hyponatremia state. The researchers will measure the volunteers' blood and urine electrolyte levels to see how these are influenced by apelin administration. As comparison, the same measurements will be done in volunteers dosed with placebo instead of apelin.

The researchers believe that apelin may be able to help to correct hyponatremia by increasing urine output. If the study focused in the healthy volunteers population is successful, the investigators will assess the effect of apelin administration in patients with chronic hyponatremia.

The study's hypothesis is that intravenous apelin will increase urinary excretion and sodium levels in healthy participants with artificially induced hyponatremia.

DETAILED DESCRIPTION:
Hyponatremia (defined as plasma sodium levels <135 mmol/l) is the most frequent electrolyte and fluid disturbance with a prevalence up to 30% in hospitalized patients. It is usually classified according to its duration, its biochemical findings (hypotonic/isotonic/hypertonic, mild/moderate/profound), its symptoms severity (mild/moderate/severe) and volume status (hypovolemic/euvolemic/hypervolemic). Chronic hyponatremia (defined as a duration > 48 hours) is associated with longer hospital stays and higher hospital costs, increased mortality and morbidity, such as gait instability, falls, osteoporosis, fractures and attention deficit. Hyponatremia is recognized as a marker of poor prognosis in multiple diseases, but the extent of its causative role has not been quantified to date. There is increasing evidence that correcting hyponatremia could improve clinical outcome.

The most common etiology of euvolemic hyponatremia is the syndrome of inappropriate antidiuresis (SIAD) which is also the main etiology of hyponatremia overall. SIAD is characterized by an imbalanced arginine vasopressin (AVP) secretion or an increased renal AVP sensitivity. This leads to free water retention, thereupon to extracellular volume expansion and a subsequent renal sodium loss resulting in hypotonic hyponatremia. Patients with SIAD are usually older adults with many comorbidities and polypharmacy making physiological studies difficult to interpret due to many possible confounders. To overcome this limitation, the investigators designed a protocol of artificial SIAD induction in healthy volunteers through administration of desmopressin and water loading.This model allowed us to develop the use of the SGLT2 inhibitors empagliflozin as a promising treatment option for SIAD.

The apelin receptor is a g-protein coupled receptor whose structure resembles the angiotensin 2 type 1 receptor. It has two endogenous ligands apelin and elabela, whose different isoforms are present in different organs and are thought to work in an autocrine/paracrine manner. Apelin is, inter alia, expressed in the magnocellular neurons of the hypothalamic supraoptic and paraventricular nuclei together with AVP and oxytocin.

Apelin has a broad spectrum of beneficial physiological effects and thus represents an attractive new target in many medical fields. For instance, it naturally displays vasodilatatory and inotropic effects and promotes glucose uptake and lipolysis. In salt and water homeostasis, apelin counteracts the effects of AVP by inhibiting central AVP release and AVP renal effect, as well as by antagonizing the vasoconstrictive effects of angiotensin II on renal afferent arterioles and increasing renal blood flow.

AVP and apelin have been shown to change in opposite directions upon hypo- and hyperosmotic challenges in healthy humans. A cross-sectional study in hyponatremic patients with SIAD or heart failure suggests that not only an increased copeptin (surrogate stoichiometric marker of AVP) but also relative insufficient apelin levels contribute to renal water reabsorption in hyponatremia. Re-establishing a physiological copeptin apelin ratio by administering exogenous apelin could therefore restore a normal salt and water balance. This concept was tested in hyponatremic rats in which an apelin-17 analog increased urine output, decreased urine osmolality and increased sodium levels to a similar extent as tolvaptan. These results suggest that apelin could become an effective treatment for SIAD, once a long-acting analog will be developed for human use. However, whether a similar effect could be induced in humans is still not known and needs to be investigated in order to characterize apelin physiology in disorders of salt and water balance.

The investigators therefore hypothesize, that the administration of intravenous [Pyr1]apelin-13, the most common apelin isoform in the blood, increases urinary excretion and thus sodium levels in healthy participants with artificially induced SIAD. In case the hypothesis is confirmed, the investigators aim to investigate the physiological effect of intravenous [Pyr1]apelin-13 administration in hyponatremic patients with chronic SIAD.

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

* Informed consent as documented by signature
* Age 18 to 65 years
* Serum sodium level 135-145mmol/l
* Clinically euvolemic status
* For female only: Due to the influence of estrogen on apelin levels, only females with combined (=containing estrogen) oral contraceptive pill will be included in order to guarantee a similar estrogen levels at each visit.

Exclusion Criteria:

* Known or suspected allergy to trial product or related products or history of multiple and/or severe allergic reaction to drugs (including study drugs) or food
* Pregnancy, wish to become pregnant during study period or breastfeeding
* Overt cardiovascular disease or abnormality in screening ECG
* Family history of sudden cardiac death or unexplained sudden death < 50 years
* Known genetic predisposition to cancer (e.g., BRCA, MEN, Lynch syndrome) or personal history/active malignant disease
* Hepatic impairment (ALAT/ASAT >3x upper limit) or liver cirrhosis
* Kidney disease (GFR < 60ml/min)
* History of epileptic seizures
* Diabetes mellitus type 1 or 2
* Other severe disease requiring regular medication intake or regular medical care
* Any daily medication (including vitamin supplements).
* Uncontrolled hypertension (systolic blood pressure >160mmHg or diastolic blood pressure >100 mmHg)
* BMI <18 or >29kg/m2
* Inability to follow the procedures of the study (e.g. due to language problems, psychological disorders, dementia).
* Participation in another study with an investigational drug within the 30 days preceding and during the present study.

Chronic SIAD patients:

Inclusion Criteria:

* Age ≥ 18 years
* Previous documented diagnosis of chronic SIAD
* Confirmed diagnosis of SIAD at screening visit defined as:

  * Plasma sodium concentration < 135 mmol/L (indirect measurement in lithium heparin plasma
  * Plasma osmolality < 300 mOsm/kg
  * Urine osmolality > 100 mOsm/kg
  * Urine sodium concentration > 30mmol/l
  * Clinical euvolemia, defined as an absence of signs of hypovolemia (orthostasis, tachycardia, decreased skin turgor, dry mucous membranes) or hypervolemia (edema, ascites)

Exclusion Criteria:

* Known or suspected allergy to trial product or related products or history of multiple and/or severe allergic reaction to drugs (including study drugs) or food.
* Pregnancy, wish to become pregnant during study period or breastfeeding
* Overt cardiovascular disease or abnormality in screening ECG
* Other potential endocrine cause of hyponatraemia:

  * Untreated glucocorticoid deficiency (Defined as morning serum cortisol levels < 300 nmol/l or serum cortisol levels < 450 nmol/l after synacthen test, in context of compatible clinical examination and medical history)
  * Untreated severe hypothyroidism (TSH > 20 mIU/L and/or free T4 < 6 pmol/L)
* Family history of sudden cardiac death or unexplained sudden death < 50 years
* Known genetic predisposition to cancer (e.g., BRCA, MEN, Lynch syndrome, …) or personal history/active malignant disease
* Hepatic impairment (ALAT/ASAT > 3x upper limit) or liver cirrhosis
* Kidney disease (GFR < 60ml/min)
* History of epileptic seizures
* Diabetes mellitus type 1 or 2
* Severe immunosuppression defined as leukocytes < 2G
* End of life care
* Severe symptomatic hyponatremia in need of treatment with 3% NaCl-solution or in need of intensive/intermediate care treatment at time of inclusion
* Risk factors for osmotic demyelination syndrome: hypokalemia (K < 3,4 mmol/L), malnutrition, advanced liver disease, alcoholism.
* Treatment with a diuretic, a SGLT2 inhibitor or a corresponding combined preparation, lithium chloride, urea, vaptans, demeclocycline or NSAIDS in the 7 days before screening (aspirin may be continued).
* Uncontrolled hypertension (systolic blood pressure > 160mmHg or diastolic blood pressure > 100 mmHg)
* BMI < 18 or > 29kg/m2
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
Total urinary excretion (ml) | assessment between timepoint 0 hours and timepoint +4 hours
  Urinary excretion, in ml, between end of water loading and one hour past study infusion completion

SECONDARY OUTCOMES:
Hourly and total urinary excretion (ml) | assessment between timepoint -2 hours and timepoint +9 hours
  Change in urine volume, in ml
Change in electrolyte free water clearance (ml/min) | assessment between timepoint -2 hours and timepoint +9 hours
  Change in electrolyte free water clearance, in ml/min
Change in free water clearance (ml/min) | assessment between timepoint -2 hours and timepoint +9 hours
  Change in free water clearance, in ml/min
Change in plasma osmolality (mOsm/kg) | assessment between baseline and timepoint +9 hours
  Change in plasma osmolality, in mOsm/kg
Change in plasma sodium (mmol/l) | assessment between baseline and timepoint +9 hours
  Change in plasma sodium, in mmol/l
Change in body weight (kg) | assessment between baseline and timepoint +9 hours
  Change in body weight, in kg

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr., Principal Investigator — University Hospital Basel; Endocrinology, Diabetes and Metabolism
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No